CLINICAL TRIAL: NCT06186752
Title: Feasibility of a Care Team-Focused Action Plan to Improve Quality of Care for Children and Adolescents With Inflammatory Bowel Disease
Brief Title: Feasibility Test of Action Planning in Pediatric IBD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-2704; R03TR004311-01A1 (NIH)
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 overall to intervention and control using permuted blocks (four) designed according to each alphabetic cluster's assigned nurse coordinator.
Who Masked: Outcomes Assessor
Masking Description: The research assistant in charge of sending out electronic surveys for data collection will be masked to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyIBD (Experimental): Each participant randomized to the intervention arm (MyIBD) will receive an individually tailored MyIBD document within a week of a scheduled outpatient clinic visit. The MyIBD document will be prepared by the patient's usual, assigned nurse coordinator together with the study's clinical champion (a nurse practitioner in the IBD program). Participants will receive a copy of the MyIBD document with language suggesting that they use it to guide decisions about care in between appointments. Each participant's primary care provider will also receive a copy of the MyIBD document. The nurse coordinator will send reminder messages to intervention-group participants (using the electronic patient portal) to access and use their MyIBD document at 1-2 months, 3-4 months, 7-8 months, and 11-12 months after initial plan creation.
  Interventions: Behavioral: MyIBD
- Usual Care (No Intervention): Each participant randomized to the control group will receive usual care in the pediatric IBD program. They will be eligible to receive a MyIBD document after completing the study (12 months after enrollment).

INTERVENTIONS:
Behavioral: MyIBD — MyIBD has two components: (1) an electronic, templated document that presents brief, actionable, tailored guidance from IBD specialists to families and other providers who care for a pediatric patient with IBD; and (2) regular, short prompts sent through the electronic patient portal to remind patients to refer to and use their MyIBD document to guide decisions about care in between appointments.
  Arms: MyIBD

SUMMARY:
The goal of this interventional study is to test the feasibility of a new communication tool, call MyIBD, in youth ages 13 to 19 years with inflammatory bowel disease. The main question[s] it aims to answer are:

* Is the MyIBD communication tool feasible to use in everyday clinical practice?
* Does the MyIBD tool have potential to improve patients' self-management skills and the quality of care they receive?

Participants who receive the MyIBD intervention will complete surveys about their care at three times points - at study enrollment, at 6 months, and at 12 months. The surveys will help the research team learn about the feasibility of using MyIBD in practice and about any effects on patients' self-management skills and quality of care.

Researchers will compare those receiving a MyIBD document to a randomly selected control group (patients receiving usual care for pediatric inflammatory bowel disease) to see if self-management skills and quality of care differ between the groups.

DETAILED DESCRIPTION:
Quality of care for youth with chronic disease suffers because of gaps in care coordination and communication among patients/families and multiple health care providers. As youth with inflammatory bowel disease (IBD) have preventive and acute care needs beyond those of peers, IBD provides an excellent use case to evaluate interventions to enhance coordination and improve quality. Electronic health records (EHRs) have unfulfilled potential to facilitate coordination and effective action among teams of providers and families. This project leverages web-based and mobile phone application access points to share patient-specific information from an IBD center's EHR. The intervention, MyIBD, has been developed with systematic input from patients, families, and providers. Our objective is to assess the feasibility of delivering tailored guidance on IBD-related health needs to families and care team members using a low-cost, low-risk health communication innovation using existing health information technology. The rationale is that brief, actionable, individually tailored guidance from IBD specialists to families and other providers will support decisions about seeking and providing timely preventive and acute care. Though the intervention builds on prior work and evidence and has been pilot tested, it requires feasibility testing in practice prior to large-scale evaluation. We will assess feasibility of MyIBD through a pilot randomized, controlled trial at one site (n=60). The study has three research aims: (1) assess the feasibility of a rollout effectiveness trial design; (2) assess the feasibility and acceptability of implementing MyIBD in a pediatric IBD clinic; (3) explore the feasibility of MyIBD to improve (a) care quality measures collected from participants and the EHR and (b) patient self-management. In Aim 1 we will assess subject recruitment, randomization, retention, intervention completion, and contamination of control subjects using a study log. For Aim 2 we will use interviews (will take place after completion of the feasibility trial) and surveys to learn about barriers and facilitators of adoption by IBD clinics and acceptability and appropriateness from the perspectives of patients/families and care providers. For Aim 3 we will use surveys and medical record data to explore change over time in family-reported care quality, patient self-management, and completion of guideline-supported quality indicators for pediatric IBD for intervention and control groups. This project is innovative in seeking to change the default ways that care team members share information and address shared responsibilities. MyIBD targets well-described barriers to coordination and incorporates behavioral strategies of individual tailoring, family participation, expert modeling, and facilitation to streamline information delivery and enhance its relevance, accessibility, and actionability. The proposed study is significant because of its potential to improve health through a low-cost intervention to enhance use of existing health information technology. The study's findings could provide a framework for EHR-supported quality improvements through learning health system research across a range of childhood-onset chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* age 13-19 years old at time of recruitment; AND
* diagnosis at least 3 months earlier of Crohn's disease, ulcerative colitis, or indeterminate colitis (to exclude families who have not had sufficient time to become familiar with condition and/or clinic personnel); AND
* receiving ongoing care at UNC (at least one visit in the past year)

Exclusion Criteria:

* speaker of a language other than English or Spanish

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of overall participants recruited and randomized | Measured and reported at the end of study year 1
  Number (0-60) will be an indicator of feasibility of implementing MyIBD in practice.
Number of intervention group participants who receive a MyIBD document | Measured and reported at the end of study year 1
  Number (0-30) of intervention-group participants who receive a MyIBD document will estimate the degree of completion of the intervention in practice.
Number of overall participants retained through baseline survey | Measured and reported at the end of study year 1
  Number (0-60) of participants who complete the baseline survey
Number of overall participants retained through 6-month survey | Measured and reported at the mid-point of study year 2
  Number (0-60) of participants who complete the 6-month survey
Number of overall participants retained through 12-month survey | Measured and reported at end of study year 2
  Number (0-60) of participants who complete the 12-month survey
Number of control group participants who receive a MyIBD document | Measured and reported at the end of study year 1
  Number (0-30) of control-group participants who (inappropriately) receive a MyIBD document is an indicator of contamination, or spreading the intervention in practice to the control group.
Number of intervention group participants who agree or completely agree that MyIBD is an acceptable intervention using the Acceptability of Intervention Measure | Reported at the end of study year 2
  Measured in the 12-month participant survey using the Acceptability of Intervention Measure (AIM), a four-item scale with five Likert-type response options from 1=Completely disagree to 5=Completely agree. Item scores are averaged to yield a scale score, with 1 indicating the lowest level of acceptability and 5 indicating the highest level.
Number of intervention group participants who agree or completely agree that MyIBD is an appropriate intervention using the Intervention Appropriateness Measure | Reported at the end of study year 2
  Measured in the 12-month participant survey using the Intervention Appropriateness Measure (IAM), a four-item scale with five Likert-type response options from 1=Completely disagree to 5=Completely agree. Item scores are averaged to yield a scale score, with 1 indicating the lowest level of appropriateness and 5 indicating the highest level.

SECONDARY OUTCOMES:
Mean self-management score on the Partners in Health scale at baseline | Measured in each participant's baseline survey; reported at end of study year 1
  Measured in the baseline participant survey using the Partners in Health Scale, a 12-item survey with 9 Likert-type response options from 0=Very Little/Never to 8=A Lot/Always. Item scores are summed to yield a total scale score from 0, indicating the lowest level of self-management skill, to 96, indicating the highest level of self-management skill.
Mean self-management score on the Partners in Health scale at 6 months | Measured in each participant's 6-month survey; reported at end of study year 2
  Measured in the 6-month participant survey using the Partners in Health Scale, a 12-item survey with 9 Likert-type response options from 0=Very Little/Never to 8=A Lot/Always. Item scores are summed to yield a total scale score from 0, indicating the lowest level of self-management skill, to 96, indicating the highest level of self-management skill.
Mean self-management score on the Partners in Health scale at 12 months | Measured in each participant's 12-month survey; reported at end of study year 2
  Measured in the 12-month participant survey using the Partners in Health Scale, a 12-item survey with 9 Likert-type response options from 0=Very Little/Never to 8=A Lot/Always. Item scores are summed to yield a total scale score from 0, indicating the lowest level of self-management skill, to 96, indicating the highest level of self-management skill.
Mean perceived Quality of Care score at baseline using the Patient Assessment of Chronic Illness Care survey | Measured in each participant's baseline survey; reported at end of study year 1
  Measured in the baseline participant survey using the Patient Assessment of Chronic Illness Care scale, a 20-item survey with 5 Likert-type responses from 1=None of the time to 5=Always. Item scores are averaged to yield an overall scale score between 1 and 5, with 1 indicating the lowest perceived care quality and 5 indicating the highest.
Mean perceived Quality of Care score at 12 months using the Patient Assessment of Chronic Illness Care survey | Measured in each participant's 12-month survey; reported at end of study year 2
  Measured in the 12-month participant survey using the Patient Assessment of Chronic Illness Care scale, a 20-item survey with 5 Likert-type responses from 1=None of the time to 5=Always. Item scores are averaged to yield an overall scale score between 1 and 5, with 1 indicating the lowest perceived care quality and 5 indicating the highest.

OTHER OUTCOMES:
Number of overall participants who completed a primary care health supervision visit in the past year, baseline | Measured by self-report in baseline survey; reported at end of study year 1
  Number (0-60) of participants who report having a primary care health supervision visit with a primary care provider in the past year
Number of overall participants who completed a primary care health supervision visit in the past year, 12 months | Measured by self-report in 12-month survey; reported at end of study year 2
  Number (0-60) of participants who report having a primary care health supervision visit with a primary care provider in the past year
Number of overall participants who completed special vaccine recommendations, baseline | Measured by self-report in baseline survey; reported at end of study year 1
  Number (0-unknown) of participants who report having completed all special vaccines recommended by IBD clinician (such as Hepatitis B booster dose, pneumococcal polysaccharide vaccine)
Number of overall participants who completed special vaccine recommendations, 12 months | Measured by self-report in 12-month survey; reported at end of study year 2
  Number (0-unknown) of participants who report having completed all special vaccines recommended by IBD clinician (such as Hepatitis B booster dose, pneumococcal polysaccharide vaccine)
Number of overall participants who participated in mood disorder screening in the past year, baseline | Measured by self-report in baseline survey; reported at end of study year 1
  Number (0-60) of participants who report participating in any mood disorder screening in the past year
Number of overall participants who participated in mood disorder screening in the past year, 12 months | Measured by self-report in 12-month survey; reported at end of study year 2
  Number (0-60) of participants who report participating in any mood disorder screening in the past year
Average number of non-injury-related visits to an emergency department (ED) in the past year, baseline | Measured by self-report in baseline survey; reported at end of study year 1
  Total count of non-injury-related ED visits by participants in the past year divided by the total number of participants
Average number of non-injury-related visits to an emergency department (ED) in the past year, 12 months | Measured by self-report in 12-month survey; reported at end of study year 2
  Total count of non-injury-related ED visits by participants in the past year divided by the total number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Neal deJong, MD, Principal Investigator — UNC-Chapel Hill School of Medicine
Locations (1):
- University of North Carolina-Chapel Hill School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become 9 to 36 months following publication and will remain available as long as the principal investigator remains actively working.
Access Criteria: See Plan Description section above for IRB or similar authorization prior to access. Once those criteria have been met, an interested investigator may contact the study PI by email (dejong@med.unc.edu); the PI would arrange for deidentified data sharing in accordance with university policy.

DOCUMENTS (1):
  • Informed Consent Form (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/52/NCT06186752/ICF_000.pdf